CLINICAL TRIAL: NCT02089724
Title: Long-term Outcome After Vemurafenib / BRAF Inhibitors Interruption in Erdheim-chester Disease
Acronym: LOVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Dr Cohen Aubart, Dr Cohen Aubart, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: medint001
Record Dates: First submitted 2014-03-15; First posted 2014-03-18 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Erdheim-Chester Disease
MeSH Terms: conditions — Erdheim-Chester Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- vemurafenib/other BRAF inhibitors

SUMMARY:
Erdheim-Chester disease (ECD) is a rare non-Langerhans cell histiocytosis. Diagnosis of ECD is based on clinical symptoms, imaging and histology with infiltration of tissues by foamy CD68 positive CD1a negative histiocytes.

Because half of the ECD patients carry a BRAFV600E mutation, we recently proposed vemurafenib, an inhibitor of mutant BRAF, as a possible targeted therapy. We have treated more than10 patients with refractory ECD with life-threatening manifestations associated with the BRAFV600E mutation and observed a short and long term efficacy.

However, vemurafenib may have several side effects and long term administration of this drug has not been evaluated. In other diseases such as melanoma, duration of administration is usually shorter, due to bad prognosis of the disease and progression despite treatment.

As in long-term follow-up, ECD patients with vemurafenib seem to have a stable disease, we want to evaluate the possibility of treatment interruption as this is what we do in our current practice. Other BRAF inhibitors, such as dabrafenib, have recently been proposed for treating BRAF mutated histiocytoses. Other BRAF inhibitor interruption treatment should also be prospectively evaluated.

DETAILED DESCRIPTION:
Erdheim-Chester disease (ECD) is a rare non-Langerhans cell histiocytosis. Diagnosis of ECD is based on clinical symptoms, imaging and histology with infiltration of tissues by foamy CD68 positive+ CD1a negative histiocytes. The clinical course mainly depends on the extent and distribution of the disease, and ranges from asymptomatic bone lesions to life-threatening manifestations. The overall mortality remains high (22% of the 100 ECD patients seen at our institution in August 2013).

Due to the rare nature of the disease (500 cases worldwide have been reported since 1930) no prospective therapeutic trial has been performed. Interferon alpha (IFN alpha), in its standard or pegylated forms, is the first line therapy for ECD. However, long-term IFN alpha treatment can lead to severe side effects. Moreover, some patients with CNS and/or cardiovascular infiltrations, the two lethal organ involvement, develop secondary resistance to high doses of IFN alpha. For refractory patients, anakinra, cladribine, tyrosine kinase inhibitors, or infliximab have been proposed as second line treatments. The optimal second line therapeutic strategy remains however to be defined, mostly because these treatments have been evaluated in only small numbers of patients.

Because half of the ECD patients carry a BRAFV600E mutation, we recently proposed vemurafenib, an inhibitor of mutant BRAF, as a possible targeted therapy. We have treated 10 patients with refractory ECD with life-threatening manifestations associated with the BRAFV600E mutation and observed a short and long term efficacy (median follow-up 9 months).

However, vemurafenib may have several side effects and long term administration of this drug has not been evaluated. In other diseases such as melanoma, duration of administration is usually shorter, due to bad prognosis of the disease and progression despite treatment.

As in long-term follow-up, ECD patients with vemurafenib seem to have a stable disease, we want to evaluate the possibility of treatment interruption as this is what we do in our current practice. Other BRAF inhibitors, such as dabrafenib, have recently been proposed for treating BRAF mutated histiocytoses.

ELIGIBILITY:
Inclusion Criteria:

* Age superior or equal to 18 years
* Clinical and radiological presentation concordant with ECD
* Presence of histological proof of ECD
* Treatment with vemurafenib or other BRAF inhibitor
* Agreement to participate

Exclusion Criteria:

* Pregnancy
* Patients who exceed the safe weight limit of the PET/CT bed (220 kg) or who cannot fit through the PET/CT bore (diameter 70 cm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population description is patients with Erdheim-Chester disease who have been treated with vemurafenib or other BRAF inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
PET scan response | 6 months (M6)
  Modification of SUVmax between M0 and M6 will be used as the main evaluation criteria for each lesion. As assessed by PERCIST criteria, patients will be classified as complete metabolic responders (CMR; complete resolution of pathologic 18F-FDG uptake), partial metabolic responders (PMR; reduction of a minimum of 30% in activity of target lesions), stable metabolic disease (SMD; not CMR, PMR, or progressive metabolic disease (PMD; increase of a minimum of 30% in activity of target lesions or presentation of a new lesion). In contrast to the PERCIST suggestions, tumor SUVmax rather than peak SUV will be measured. Target lesion will be defined by the most active lesion on FDG-PET/CT study before treatment and, for each patient, one or two secondary target lesions among the most active lesions will also be studied. Side-by-side image review and analysis will be performed to ascertain that the SUVmax is derived from the same lesions on baseline and follow-up scans

SECONDARY OUTCOMES:
Specific organ assessment (cardiac, retroperitoneal, neurological) | Months 6 and Months 12
PET scan | Months 12
CRp value (mg/liter) | Months 6 and Months 12

CONTACTS AND LOCATIONS:
Overall Officials: Julien Haroche, MD, PhD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière; Fleur Cohen Aubart, MD, PhD, Study Director — Groupe Hospitalier Pitié-Salpêtrière; Eli L. Diamond, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- AP-HP, Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Background] Haroche J, Arnaud L, Cohen-Aubart F, Hervier B, Charlotte F, Emile JF, Amoura Z. Erdheim-Chester disease. Curr Rheumatol Rep. 2014 Apr;16(4):412. doi: 10.1007/s11926-014-0412-0. PMID 24532298
- [Background] Haroche J, Cohen-Aubart F, Emile JF, Arnaud L, Maksud P, Charlotte F, Cluzel P, Drier A, Hervier B, Benameur N, Besnard S, Donadieu J, Amoura Z. Dramatic efficacy of vemurafenib in both multisystemic and refractory Erdheim-Chester disease and Langerhans cell histiocytosis harboring the BRAF V600E mutation. Blood. 2013 Feb 28;121(9):1495-500. doi: 10.1182/blood-2012-07-446286. Epub 2012 Dec 20. PMID 23258922
- [Background] Haroche J, Charlotte F, Arnaud L, von Deimling A, Helias-Rodzewicz Z, Hervier B, Cohen-Aubart F, Launay D, Lesot A, Mokhtari K, Canioni D, Galmiche L, Rose C, Schmalzing M, Croockewit S, Kambouchner M, Copin MC, Fraitag S, Sahm F, Brousse N, Amoura Z, Donadieu J, Emile JF. High prevalence of BRAF V600E mutations in Erdheim-Chester disease but not in other non-Langerhans cell histiocytoses. Blood. 2012 Sep 27;120(13):2700-3. doi: 10.1182/blood-2012-05-430140. Epub 2012 Aug 9. PMID 22879539